CLINICAL TRIAL: NCT00759317
Title: Physiologic Monitoring of Antidepressant Medication Effects in Normal Controls Subjects I
Brief Title: Physiologic Monitoring of Antidepressant Treatment Response
Acronym: Ven Nls I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Ven Nls I
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Depression
Keywords: normal controls
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): venlafaxine
  Interventions: Drug: venlafaxine (Effexor)
- 2 (Placebo Comparator)
  Interventions: Drug: venlafaxine (Effexor)

INTERVENTIONS:
Drug: venlafaxine (Effexor) — Matching capsules containing either venlafaxine 37.5 mg. or placebo will be prepared by the UCLA Pharmacy for the initial phase of the study. For the open-label phase of the study, subjects will receive the medication and dosage that is clinically indicated by the subject's primary physician in the community. After a one-week placebo lead-in, subjects will be randomly assigned to receive one capsule of either venlafaxine or placebo, with the dosage increase every two days until subjects receive four capsules daily (subjects will achieve a dose 150 mg. of venlafaxine after 7 days). The first dose will be administered in the morning, with subsequent capsules added on a b.i.d. schedule.

SUMMARY:
Study Objectives:

* to identify neurophysiologic effects of venlafaxine treatment in normal controls using quantitative EEG (QEEG) cordance
* to examine the effects of venlafaxine on different rating scales measuring mood and anxiety (e.g., Ham-D, BDI, SCL-90, POMS-BI, Visual Analog Mood Scale, SSRS, SASS, Q-LES-Q and SF-36) as well as on measures of cognitive and psychosocial function (i.e., Stroop, PASAT, RAVLT, Trailmaking A and B, Digit-Symbol, Grooved Pegboard, Multidimensional Health Locus of Control, Temperament and Character Inventory, Interpersonal Support Evaluation List, Godin Leisure-Time Questionnaire, and Pittsburgh Sleep Quality Index) in normal control subjects, and the association of changes in cordance with changes in thinking and memory.
* to identify physiologic effects of venlafaxine treatment in normal controls using heart rate and immune function measures

DETAILED DESCRIPTION:
Pilot data suggest that in depressed patients treated with fluoxetine or venlafaxine, QEEG cordance detects changes of brain function within individual subjects as soon as two days after initiation of treatment. Changes in cordance appear to be specific (i.e., do not occur in the absence of clinical improvement), and frequently precede examiner ratings of improvement (Leuchter et al., 1997; Cook et al., in submission). In addition, patterns of cordance at baseline may indicate which patients are most likely to respond to fluoxetine or venlafaxine treatment (Cook et al., 1999).

Findings using cordance contrast with those reported in previous QEEG studies of antidepressant medications, performed in depressed as well as normal control subjects. These studies have shown QEEG effects of antidepressant medication, such as decreased theta or alpha band activity, that are not related to changes in clinical state. In particular, normal subjects receiving antidepressant medications have been reported to show changes in conventional QEEG power measurements that may be useful characteristics of antidepressant medication for medication development purposes. Similar changes in QEEG power have been reported in depressed subjects who do not show clinical improvement (Saletu et al 1982, 1983, 1985, 1986, 1987, 1988; Sannita et al 1983, 1990; Itil et al 1984; Herrmann et al., 1991; Luthringer et al., 1996). The relationship of these immediate EEG changes in control subjects to eventual clinical response in a depressed population is unclear. Other QEEG work with depressed subjects has found that changes from baseline in theta power early in the course of treatment may characterize groups of depressed patients who are more likely to respond to antidepressant treatment (Ulrich et al., 1994). Unfortunately, the changes lacked the specificity to allow response prediction for individual subjects, and the physiologic meaning of these changes in theta power is not clear.

We previously have shown that absolute and relative power are complementary measures of brain activity (Leuchter et al., 1993). Cordance is a new QEEG measure that combines information from both absolute and relative power measures (Leuchter et al., 1994). In validation against data collected simultaneously with 15O positron emission tomography (PET), cordance values in the theta frequency band (4-8 Hz) were found to be positively correlated with cortical perfusion, and this correlation was stronger than that between perfusion and either absolute or relative theta power (Leuchter et al., 1999). The correlation of cordance with regional cortical perfusion provides a physiologic context in which to interpret this measure.

In a series of depressed subjects receiving open-label treatment, we previously have shown that cordance detects changes in prefrontal activity (using a within-subjects design) as early as after three days of treatment in patients who will later show clinical response to antidepressant medication. Subjects who did not respond to antidepressant medication, as well as those receiving placebo, did not show these early changes in cordance (Leuchter et al 1997; Cook et al 1998; Cook et al., in submission). These data suggest that QEEG cordance may be a more specific indicator of antidepressant treatment effectiveness than traditional QEEG power measures, since antidepressant non-responders and placebo treated subjects showed no early change in this measure. It is important, however, to determine if the effects that we have observed in depressed subjects during treatment are specific for this population, or are seen in normal controls as well. First, examination of specificity in normal controls during treatment is a logical first step in the process of examining other groups, eventually including other patient groups. Second, examination of normal subjects will help us to determine whether the observed changes in brain function are a pharmacodynamic effect of antidepressant medication which could be seen in any individual, or an effect seen exclusively in depressed subjects early in the course of effective antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be between the ages of 18 - 65 and in good health (i.e., free of any medical condition known to affect brain function).

Exclusion Criteria:

* All subjects will have no serious medical illness such as high blood pressure, heart disease, renal impairment, or cirrhosis of the liver. This will be assured by making sure that prospective subjects have had a normal physical exam with in one year prior to entry of the study.
* The investigators will also exclude subjects who meet DSM-IV axis I criteria for a mood, anxiety, cognitive, or psychotic disorder on the basis of a SCID-P interview, as well as those meeting criteria for cluster A or B axis II diagnoses.
* Subjects with a history of current or past active suicidal ideation or suicide attempts will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-06; Primary Completion 2002-08 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Laboratory of Brain, Behavior, and Pharmacology, Los Angeles, California, United States

REFERENCES:
- [Background] Hunter AM, Cook IA, Abrams M, Leuchter AF. Neurophysiologic effects of repeated exposure to antidepressant medication: are brain functional changes during antidepressant administration influenced by learning processes? Med Hypotheses. 2013 Dec;81(6):1004-11. doi: 10.1016/j.mehy.2013.09.016. Epub 2013 Sep 17. PMID 24112999
- [Result] Leuchter AF, Cook IA, Hunter AM, Cai C, Horvath S. Resting-state quantitative electroencephalography reveals increased neurophysiologic connectivity in depression. PLoS One. 2012;7(2):e32508. doi: 10.1371/journal.pone.0032508. Epub 2012 Feb 24. PMID 22384265